CLINICAL TRIAL: NCT07301840
Title: Ultrasound-guided Erector Spinae Plane Block Versus Local Wound Infiltration in Breast Conservative Surgery, Randomized Double Blinded Comparative Study
Brief Title: Ultrasound-guided Erector Spinae Plane Block Versus Local Wound Infiltration in Breast Conservative Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tasneem Hassan El-Tohamy, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-433-2024
Record Dates: First submitted 2025-11-13; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Local Wound Infiltration; Erector Spina Plan Block; Nerve Block/Methods; Post Operative Analgesia; Pain Management
Keywords: Erector Spinae Plane Block; Local wound infiltration; Postoperative analgesia; Breast conservative surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized Double Blinded Comparative Study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (experimental group): will receive US guided ESPB (Experimental)
  Interventions: Procedure: Erector Spinae Plane Block
- Group 2 (controlled group): will receive local wound infiltration (Active Comparator)
  Interventions: Procedure: Local Wound Infiltration

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Typical ESPB
  Arms: Group 1 (experimental group): will receive US guided ESPB
Procedure: Local Wound Infiltration — Preemptive Local Wound Infiltration
  Arms: Group 2 (controlled group): will receive local wound infiltration

SUMMARY:
Abstract

Background:

Postoperative pain management is a crucial component of patient care following breast conservative surgery. This study compares the efficacy of ultrasound-guided Erector Spinae Plane Block (ESPB) and Local Wound Infiltration (LWI) in managing acute postoperative pain in these surgeries.

Objectives:

This randomized, double-blinded, controlled clinical trial aims to compare the analgesic efficacy and safety of ultrasound-guided ESPB and LWI in patients undergoing breast conservative surgery.

Patients and methods:

Adult female patients (aged 18-75, ASA II) scheduled for breast conservative surgery were randomly assigned to either the ESPB or LWI group. The primary outcome was total morphine consumption in the first 24 hours postoperatively. Secondary outcomes included; intraoperative fentanyl consumption, hemodynamic parameters (mean arterial blood pressure and heart rate), time of first rescue analgesia, postoperative pain scores, the incidence of postoperative nausea and vomiting (PONV) and patient satisfaction. Complications such as local anesthetic toxicity and respiratory depression were also assessed.

Key Words:

Erector Spinae Plane Block (ESPB), Local wound infiltration, Postoperative analgesia, Breast conservative surgery

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* Genders eligible for study: females.
* ASA II.
* Patients scheduled for breast conservative surgery.
* Ability to provide informed consent or, if unable, consent obtained from a legal representative

Exclusion Criteria:

* Patient refusal.
* Inability to provide informed consent.
* ASA III-IV.
* Known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).
* Pregnant or lactating women.
* History of psychological disorders and/or chronic pain. 25
* Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.
* Male patients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Total amount of morphine consumed postoperatively for 24 hours. | up to 24 hours postoperative
  Total amount of morphine consumed postoperatively for 24 hours (mg/kg)

SECONDARY OUTCOMES:
Total amount of fentanyl consumed intraoperatively | Perioperative/Periprocedural
  Total amount of fentanyl consumed intraoperatively (mic/kg)
Hemodynamics: heart rate intraoperatively at 30-minute intervals in comparison to baseline readings. | Perioperative/Periprocedural
  Hemodynamics: heart rate intraoperatively at 30-minute intervals in comparison to baseline readings (beats/min)
Hemodynamics: mean arterial blood pressure intraoperatively at 30-minute intervals in comparison to baseline readings. | Perioperative/Periprocedural
  Hemodynamics: mean arterial blood pressure intraoperatively at 30-minute intervals in comparison to baseline readings (mmHg)
Heart rate at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively. | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively.
  Heart rate at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively (beats/min)
Mean arterial blood pressure at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively. | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively.
  Mean arterial blood pressure at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively (mmHg)
The visual analog scale (VAS) (at rest and during movement) at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively. | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively.
  The visual analog scale (VAS) is a pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10cm)
Postoperative nausea and vomiting (PONV) as side effects of morphine. | up to 24 hours postoperative
  Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe=vomiting >one attack).
Time of first rescue analgesia intra-operative (Fentanyl) | up to 24 hours postoperative
  Time of first rescue analgesia (min)
Time of first rescue analgesia post-operative (Morphine) | up to 24 hours postoperative
  Time of first rescue analgesia (hrs.)
Complications such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture. (US check postoperative). | up to 24 hours postoperative
  Complications such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture. (US check postoperative).
Morphine related complications such as respiratory depression, urine retention or pruritic | up to 24 hours postoperative
  Morphine related complications such as respiratory depression, urine retention or pruritic
Patient satisfaction the patient will be classified in this group into satisfied or not. | up to 24 hours postoperative
  Patient satisfaction the patient will be classified in this group into satisfied or not.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes